CLINICAL TRIAL: NCT01358591
Title: Effect of a High Calcium Breakfast on Exercise Metabolism and Appetite
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Northumbria University (Other)
Responsible Party: Principal Investigator, Javier Gonzalez, PhD Student, Northumbria University
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: 32AN1
Record Dates: First submitted 2011-05-20; First posted 2011-05-23 (Estimated); Last update posted 2012-06-05 (Estimated); Status verified 2012-06

CONDITIONS: Exercise Fat Oxidation

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- Control Breakfast (Sham Comparator): Normal calcium breakfast.
  Interventions: Dietary Supplement: Control
- High calcium breakfast (Experimental): High calcium breakfast.
  Interventions: Dietary Supplement: High calcium milk

INTERVENTIONS:
Dietary Supplement: High calcium milk — High calcium milk (9 mg/kgBM)
  Arms: High calcium breakfast
Dietary Supplement: Control — Regular Milk
  Arms: Control Breakfast

SUMMARY:
The purpose of this study is to assess the effect of a high calcium breakfast on substrate metabolism during exercise and appetite throughout the day.

ELIGIBILITY:
Inclusion Criteria:

* Male
* Aged 18-45 years
* Physically active - able to run continuously for 1 h.

Exclusion Criteria:

* Smokers
* Food Allergies
* Metabolic Disorders
* Consuming herbal/dietary supplements
* Gastric Problems

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 9 (Actual)
Dates: Start 2011-05; Primary Completion 2011-11 (Actual); Study Completion 2011-11 (Actual)

PRIMARY OUTCOMES:
Total fat oxidised during 60 min of exercise (g). | 1 hour
  Assessed by indirect calorimetry

SECONDARY OUTCOMES:
Blood glucose concentration | 2 hour
  2 h incremental area under the curve for blood glucose following breakfast consumption
Serum Insulin Concentration | 2 hour
  2 h area under the curve for serum insulin following breakfast consumption
Subjective appetite ratings | 3 hour
  Subjective ratings of appetite assessed by visual analogue scales.

CONTACTS AND LOCATIONS:
Locations (1):
- Northumbria University, Newcastle upon Tyne, Tyne and Wear, United Kingdom